CLINICAL TRIAL: NCT05296902
Title: Single Center Open-Label Post Market Clinical Follow-Up (PMCF) -Study on the Performance of Safety of SILKAM® Suture Material in Oral Surgery
Brief Title: Performance of Safety of SILKAM® Suture Material in Oral Surgery
Acronym: SILKOS
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2038
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Tooth, Impacted; Teeth Impact; Tooth Impaction; Mucosal Wound
Keywords: Tooth distraction; Removal of impacted Teeth; Oral Surgery; Dental Implant; Observational Study
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SILKAM®: SILKAM® is a non-absorbable sterile suture material made from braided silk fibrils. It is available either undyed (white) or dyed black with hematein and is coated with refined paraffin wax or beeswax.
  Interventions: Device: Mucosal Closure

INTERVENTIONS:
Device: Mucosal Closure — mucosal closure in oral surgery (mucosal sutures)

SUMMARY:
Assessment of SILKAM® suture material in mucosal closure in oral surgery (mucosal sutures). A prospective, monocentric, single arm observational study.

DETAILED DESCRIPTION:
The aim of this Non Interventional Study is to collect systematically and proactively different clinical parameters regarding safety, effectiveness, and performance of SILKAM® suture material under the daily routine clinical practice when is intended to be used for oral surgery. All patients enrolled will be prospectively followed until suture removal, which takes place approximately one week post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mucosal wound closure using SILKAM® as suture material in oral surgery (in the event that more than one incision is performed in the same patient, only one incision will be considered).

Exclusion Criteria:

* Patients taking medication that might affect wound healing
* Patients having a condition that might affect wound healing.
* Patients with hypersensitivity or allergy to the suture material.
* Participation in another (Randomized) Clinical Trial / Clinical Study.
* Non-compliance of patient (i.e. dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing mucosal closure in oral surgery (mucosal sutures).
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Surgical Wound Dehiscence rate | until day of suture removal (approximately 1 week after surgery)
  Pathologic process consisting of a partial or complete disruption of the layers of a surgical wound.
Complication rate | until day of suture removal (approximately 1 week after surgery)
  Complications rate according to the "Classification of Askar" as Grade 1 (Localized complication(s) accompanied by no adverse effects on the success of the surgery) and Grade 2 (Localized complication(s) accompanied by adverse effects on the success of the surgery).

SECONDARY OUTCOMES:
Complication rate | until day of suture removal (approximately 1 week after surgery)
  Complications rate according to the "Classification of Askar" as Grade 3 (Localized or systemic complication(s) that impairs the patient's daily routine but does not require hospitalization), Grade 4 (Localized or systemic complication(s) that impairs the patient's daily routine and requires hospitalization), Grade 5 (Localized or systemic complication(s) that inflicts irreversible damage to >1 anatomical structures), or Grade 6 (Localized or systemic complication(s) that lead to death.
Pain assessment using the visual analogue scale (VAS 1-100) | until day of suture removal (approximately 1 week after surgery)
  This parameter will be noted according to the Patient self assessment using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal pain".
Satisfaction of the patient using the visual analogue scale (VAS 1-100) | until day of suture removal (approximately 1 week after surgery)
  This parameter will be noted according to the Patient self assessment using the Visual Analogue Scale (VAS) which state "0" at one end representing "completely satisfied" and "100" at the opposite end representing "not at all satisfied".
Wound healing assessment using the visual analogue scale (VAS 1-100) | until day of suture removal (approximately 1 week after surgery)
  This parameter will be noted by the surgeon using the Visual Analogue Scale (VAS) which state "0" at one end representing "very good wound healing" and "100" at the opposite end representing "very bad wound healing".
Assessment of the handling of the suture material | intraoperatively
  Evaluation of the handling of the suture material in five categories (Knot security, Knot run down, Knot pull tensile strength, Tissue drag, Pliability) with the 5 evaluation levels each: 'excellent', 'very good', 'good', 'satisfied' and 'poor' transferred into the evaluation scores 5, 4, 3, 2 and 1.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Quevedo Pou, Dr., Principal Investigator — Facultat D'odontologia. Universitat Internacional de Catalunya
Locations (1):
- Facultat D'odontologia. Universitat Internacional de Catalunya, Sant Cugat del Vallès, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No